CLINICAL TRIAL: NCT06483737
Title: Human Albumin Infusion in Liver Cirrhosis and Overt Hepatic Encephalopathy (HACHE): an Invesitgator-initiated, Open-label, Multicenter, Randomized Controlled Trial
Brief Title: Human Albumin Infusion in Liver Cirrhosis and Overt Hepatic Encephalopathy (HACHE)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Xingshun Qi, Director of Department of Gastroenterology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XHNKKY-OHE-RCT
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Overt Hepatic Encephalopathy
Keywords: hepatic encephalopathy; liver cirrhosis; human albumin; inflammation; oxidative stress; survival
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis; Inflammation | interventions — Albumins; Lactulose; Rifaximin; ornithylaspartate; Amino Acids, Branched-Chain; Arginine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Modified dosage group (Experimental): Intravenous infusion of human albumin 30-60g.
  Interventions: Drug: Human albumin infusion at a modified dosage; Drug: Lactulose; Drug: Rifaximin; Drug: Ornithine Aspartate; Drug: Branched-Chain Amino Acids; Drug: Arginine
- Routine dosage group (Active Comparator): Intravenous infusion of human albumin 10-20g.
  Interventions: Drug: Human albumin infusion at a routine dosage; Drug: Lactulose; Drug: Rifaximin; Drug: Ornithine Aspartate; Drug: Branched-Chain Amino Acids; Drug: Arginine

INTERVENTIONS:
Drug: Human albumin infusion at a modified dosage — Participants receive intravenous infusion of human albumin at different dosages according to the serum albumin level.
  Other Names: AlbuRx
  Arms: Modified dosage group
Drug: Human albumin infusion at a routine dosage — Participants receive intravenous infusion of human albumin according to the current clinical practice.
  Other Names: AlbuRx
  Arms: Routine dosage group
Drug: Lactulose — All participants will receive standard treatment of overt HE according to the current practice guideline.
  Other Names: Duphalac
Drug: Rifaximin — All participants will receive standard treatment of overt HE according to the current practice guideline.
  Other Names: Xifaxan
Drug: Ornithine Aspartate — All participants will receive standard treatment of overt HE according to the current practice guideline.
Drug: Branched-Chain Amino Acids — All participants will receive standard treatment of overt HE according to the current practice guideline.
  Other Names: Compound amino acid injection
Drug: Arginine — All participants will receive standard treatment of overt HE according to the current practice guideline.
  Other Names: Arginine Hydrochloride Injection

SUMMARY:
Hepatic encephalopathy (HE), a severe complication of decompensated cirrhosis, is characterized as neurocognitive dysfunction. Emerging evidence suggests the potential role of human albumin infusion for the treatment of HE, but its optimal dosage remains undefined. Therefore, the investigators planned a randomized controlled trial (RCT) to compare the efficacy of human albumin infusion at different dosages in in patients with liver cirrhosis and overt HE.

DETAILED DESCRIPTION:
Overall, 174 patients with a diagnosis of liver cirrhosis, overt HE, and a serum albumin level of 23-30g/L will be enrolled. They will be stratified according to the severity of overt HE and randomly assigned at a ratio of 1:1 into the groups of human albumin infusion at a modified dosage and a routine dosage. The primary endpoint is the improvement of overt HE within 3-5 days after treatment. The secondary endpoints include recurrence of overt HE, survival, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* A definite diagnosis of liver cirrhosis and overt HE
* A serum albumin level of 23-30g/L
* Age ≥18 years old
* Sign the informed consent

Exclusion Criteria:

* Contraindications to human albumin infusion
* A history of transjugular intrahepatic portosystemic shunt
* A diagnosis of acute liver failure
* Severe heart and/or lung diseases
* Psychiatric or nervous diseases
* Pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of overt HE. | 3-5 days
  The change of HE is defined as a decrease or an increase of at least one grade of the West Haven criteria after treatment.

SECONDARY OUTCOMES:
Reversal of overt HE. | 3-5 days
  The reversal of HE is defined as clinical symptoms of overt HE disappear after treatment.
Recurrence of overt HE. | 3 months
  Clinical symptoms related to overt HE recur and can be diagnosed with overt HE again according to the West Haven criteria.
Adverse events | 3 months
  Adverse events will be monitored, including allergy, heart failure, pulmonary edema, acute hemolysis, renal dysfunction, and neuropsychiatric abnormalities.
Survival | 3 months
  All participants will be followed by telephone to record survival status, including the major cause and date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Xingshun Qi, Principal Investigator — Department of Gastroenterology, General Hospital of Northern Theater Command
Locations (1):
- Department of Gastroenterology, General Hospital of Northern Theater Command (formerly called General Hospital of Shenyang Military Area), Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma BC, Singh J, Srivastava S, Sangam A, Mantri AK, Trehanpati N, Sarin SK. Randomized controlled trial comparing lactulose plus albumin versus lactulose alone for treatment of hepatic encephalopathy. J Gastroenterol Hepatol. 2017 Jun;32(6):1234-1239. doi: 10.1111/jgh.13666. PMID 27885712
- [Background] Simon-Talero M, Garcia-Martinez R, Torrens M, Augustin S, Gomez S, Pereira G, Guevara M, Gines P, Soriano G, Roman E, Sanchez-Delgado J, Ferrer R, Nieto JC, Sunye P, Fuentes I, Esteban R, Cordoba J. Effects of intravenous albumin in patients with cirrhosis and episodic hepatic encephalopathy: a randomized double-blind study. J Hepatol. 2013 Dec;59(6):1184-92. doi: 10.1016/j.jhep.2013.07.020. Epub 2013 Jul 19. PMID 23872605
- [Background] China L, Freemantle N, Forrest E, Kallis Y, Ryder SD, Wright G, Portal AJ, Becares Salles N, Gilroy DW, O'Brien A; ATTIRE Trial Investigators. A Randomized Trial of Albumin Infusions in Hospitalized Patients with Cirrhosis. N Engl J Med. 2021 Mar 4;384(9):808-817. doi: 10.1056/NEJMoa2022166. PMID 33657293
- [Background] Bai Z, Bernardi M, Yoshida EM, Li H, Guo X, Mendez-Sanchez N, Li Y, Wang R, Deng J, Qi X. Albumin infusion may decrease the incidence and severity of overt hepatic encephalopathy in liver cirrhosis. Aging (Albany NY). 2019 Oct 8;11(19):8502-8525. doi: 10.18632/aging.102335. Epub 2019 Oct 8. PMID 31596729
- [Background] Bai Z, Mendez-Sanchez N, Romeiro FG, Mancuso A, Philips CA, Tacke F, Basaranoglu M, Primignani M, Ibrahim M, Wong YJ, Nery FG, Teschke R, Ferreira CN, Munoz AE, Pinyopornpanish K, Thevenot T, Singh SP, Mohanty A, Satapathy SK, Ridola L, Maruyama H, Cholongitas E, Levi Sandri GB, Yang L, Shalimar, Yang Y, Villa E, Krag A, Wong F, Jalan R, O'Brien A, Bernardi M, Qi X; Liver Cirrhosis-related Complications (LCC)-International Special Interest Group. Use of albumin infusion for cirrhosis-related complications: An international position statement. JHEP Rep. 2023 May 5;5(8):100785. doi: 10.1016/j.jhepr.2023.100785. eCollection 2023 Aug. PMID 37456673
- [Derived] Li Q, Tong H, Liu X, Liao F, Ma H, Zhou Z, Liu F, Shi H, Wang Z, Sun Y, Yao Q, Feng Y, Li X, Feng J, He Z, Peng Y, Bai Z, Zhu R, Cheng D, Xu C, He S, Yu H, Xie C, Yuan J, Wang X, Yang H, Zou Y, Li S, Li T, Hu S, Chen C, Chen Z, Lantinga MA, Bernardi M, Qi X, Tang C; On the behalf of Young Member Group of Chinese Gastroenterology Society. Human Albumin infusion in liver Cirrhosis and overt Hepatic Encephalopathy (HACHE): protocol of an investigator-initiated, open-label, multicentre, randomised controlled trial. BMJ Open. 2025 Nov 5;15(11):e094300. doi: 10.1136/bmjopen-2024-094300. PMID 41198206